CLINICAL TRIAL: NCT00747773
Title: A Study Of Cryospray Ablationtm Using Surgical Resection Specimens To Determine Safety And Histological Effect In The Lung
Brief Title: Cryospray Ablation of Surgical Resection Specimens To Determine Safety And Histological Effect In The Lung
Acronym: CSAir 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00008-00
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; CryoPsray Ablation; CSA therapy; CSA treatment; Lobectomy; lung resection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CryoSpray Ablation System — CSA Medical, Inc. (formerly CryMed Technologies, Inc.) received FDA market clearance for the CSA System (CryoSpray AblationTM System, formally Cryo Ablator System) on April 21, 2006. It is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications" (K070893). As defined by the FDA, the CSA System is a cryosurgical unit with a liquid nitrogen cooled cryocatheter and accessories used to destroy tissue during surgical procedures by applying extreme cold

SUMMARY:
The purpose of this study is to evaluate the feasibility and general safety in the human airway as well as assess the safety and depth and area of treatment using liquid nitrogen sprayed through a catheter via flexible fiber optic bronchoscopy (FFB) using surgical resection specimens from patients undergoing lobectomy.

DETAILED DESCRIPTION:
The primary endpoints for this study are patient safety and the histological effects of cryospray therapy in lobectomy patients.

The proposed study is a single center study to evaluate the safety and treatment effect of sprayed liquid nitrogen through a catheter via FFB using surgical resection specimens from patients undergoing lobectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age
* Lobectomy planned based on clinical situation not related to this study.
* Deemed operable based on institutional criteria.

Exclusion Criteria:

* Pregnant or nursing
* Planning to sire a child while enrolled in the study
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.
* Refusal or inability to give consent.
* Concurrent chemotherapy.
* Prior radiation therapy which involved the lungs
* Medical contraindication or potential problem that would preclude study participation
* Concurrent participation in other experimental studies
* Uncontrolled coagulopathy or bleeding diathesis
* Serious medical illness, including:
* Uncontrolled congestive heart failure
* Uncontrolled angina
* Myocardial infarction
* Cerebrovascular accident within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint for this study is patient safety | Throughout study
The primary efficay endpoint is histological effects of cryospray therapy in lobectomy patients | Throughout Study

CONTACTS AND LOCATIONS:
Overall Officials: Willaim Krimsky, MD, Principal Investigator — PCCAB, Franklin Square Hospital Center
Locations (1):
- Franklin Square Hospital Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Krimsky WS, Broussard JN, Sarkar SA, Harley DP. Bronchoscopic spray cryotherapy: assessment of safety and depth of airway injury. J Thorac Cardiovasc Surg. 2010 Mar;139(3):781-2. doi: 10.1016/j.jtcvs.2009.03.051. Epub 2009 Aug 6. No abstract available. PMID 19664781